CLINICAL TRIAL: NCT02905890
Title: Hormonal Contraception and Bacterial Vaginosis (HCBV): The Effect of Norethisterone Enanthate on Recurrent Bacterial Vaginosis Among Women at High Risk for HIV Infection in Kampala, Uganda
Brief Title: The Effect of Norethisterone Enanthate on Recurrent Bacterial Vaginosis
Acronym: HCBV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Imperial College London (Other); University of Liverpool (Other); MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QA906
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Bacterial Vaginosis; HIV
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — norethindrone enanthate; Condoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norethisterone enanthate plus condoms (Experimental): 200 mg Norethisterone enanthate intramuscularly every eight weeks at enrolment, 2 and 4 months. Counseling and condoms will be provided at enrolment, 1, 2, 3 and 4 months.
  Interventions: Drug: Norethisterone enantate; Device: Condoms
- Condoms only (Active Comparator): Counseling and condoms will be provided at enrolment, 1, 2, 3 and 4 months.
  Interventions: Device: Condoms

INTERVENTIONS:
Drug: Norethisterone enantate — Noristerat® 200mg, solution for intramuscular injection given every 8 weeks
  Other Names: Noristerat
  Arms: Norethisterone enanthate plus condoms
Device: Condoms — Latex male condoms

SUMMARY:
The proposed study, Hormonal Contraception & BV (HCBV), will investigate the effect of NET-EN and DMPA on recurrent BV, vaginal microbiota and inflammatory markers among women at high risk for HIV in Kampala, Uganda. The hypothesis is that NET-EN will show a similar beneficial effect on recurrent BV and vaginal microbiota as DMPA, without inducing signs of mucosal inflammation.

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) is highly prevalent among women in Africa and is associated with HIV acquisition. BV has been described as a dysbiosis, or a microbial imbalance, and is treated with metronidazole; however, once treated, it often recurs rapidly. Developing robust treatment strategies to prevent recurrent BV is important for HIV prevention in key populations at high risk for HIV infection.

There is evidence that hormonal contraceptives, including depot medroxyprogesterone acetate (DMPA), decrease BV recurrence; however, there is also evidence that DMPA increases the risk of HIV infection. Encouraging women to start or switch to an alternative progestin injectable such as norethisterone enantate (NET-EN) may mitigate HIV risk whilst decreasing the risk of recurrent BV. To date, there are no published studies that have investigated the effect of NET-EN on vaginal microbiota.

The proposed study will investigate the effect of NET-EN and DMPA on recurrent BV, vaginal microbiota and inflammatory markers among women at high risk for HIV in the Good Health for Women Project in Kampala, Uganda. Consenting and eligible women will be treated for BV, and randomised to either NET-EN plus condoms or condoms only. Women currently using DMPA will be enrolled as an observational comparison arm. All participants will be interviewed and examined; samples for vaginal microbiota, sexually transmitted infections, and inflammatory markers will be obtained. Women will be followed up after 1 week, and 1, 2, 3, 4 and 6 months. The primary outcomes will be differences in vaginal microbiota clusters, time to recurrent BV, and inflammatory markers. Qualitative research will be carried out to assess the acceptability of, and adherence to, NET-EN.

ELIGIBILITY:
Inclusion Criteria:

* BV positive by Nugent score
* HIV negative
* Capable of providing written informed consent

Exclusion Criteria:

* Currently pregnant or using a reliable contraception (e.g. injectables, intrauterine devices, implant, oral contraceptive pills)
* Desiring pregnancy in the next year
* History of tubal ligation or hysterectomy
* Contraindication to progestin-only contraceptives
* Unable to comprehend consent material because of language barrier or psychological difficulty

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Time to diagnosis of recurrent BV | 6 months

SECONDARY OUTCOMES:
Proportional of participants with Lactobacillus-dominant cluster | 6 months
Concentration of markers for inflammation | 6 months
  Twenty-four soluble immune proteins will be quantified by in-house multiplex bead immunoassay including interleukin(IL)-1α, IL1β, IL-2, IL4, IL-6, IL-7, IL- 8, IL-12, IL-15, IL16, IFN-g, MIP-1β, SDF1β, TNF-α, IP-10, RANTES, GM-CSF, G-CSF, MIG, IFN- -β, TGF-β, MCP-1, MCP-2, MIP-3α and other immune proteins as appropriate.
Acceptability of norethisterone enanthate as measured by qualitative interviews | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna C Francis, MSc MPH PHD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- MRC/UVRI Mengo Clinic and Research Station, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data from consenting participants will be made available to third parties in line with Open Access data requirements after a period of exclusive use by the study investigators

REFERENCES:
- [Background] Mitchell C, Marrazzo J. Bacterial vaginosis and the cervicovaginal immune response. Am J Reprod Immunol. 2014 Jun;71(6):555-63. doi: 10.1111/aji.12264. PMID 24832618
- [Background] Bradshaw CS, Morton AN, Hocking J, Garland SM, Morris MB, Moss LM, Horvath LB, Kuzevska I, Fairley CK. High recurrence rates of bacterial vaginosis over the course of 12 months after oral metronidazole therapy and factors associated with recurrence. J Infect Dis. 2006 Jun 1;193(11):1478-86. doi: 10.1086/503780. Epub 2006 Apr 26. PMID 16652274
- [Background] Francis SC, Looker C, Vandepitte J, Bukenya J, Mayanja Y, Nakubulwa S, Hughes P, Hayes RJ, Weiss HA, Grosskurth H. Bacterial vaginosis among women at high risk for HIV in Uganda: high rate of recurrent diagnosis despite treatment. Sex Transm Infect. 2016 Mar;92(2):142-8. doi: 10.1136/sextrans-2015-052160. Epub 2015 Aug 7. PMID 26253744
- [Background] Vodstrcil LA, Hocking JS, Law M, Walker S, Tabrizi SN, Fairley CK, Bradshaw CS. Hormonal contraception is associated with a reduced risk of bacterial vaginosis: a systematic review and meta-analysis. PLoS One. 2013 Sep 4;8(9):e73055. doi: 10.1371/journal.pone.0073055. eCollection 2013. PMID 24023807
- [Background] Bradshaw CS, Brotman RM. Making inroads into improving treatment of bacterial vaginosis - striving for long-term cure. BMC Infect Dis. 2015 Jul 29;15:292. doi: 10.1186/s12879-015-1027-4. PMID 26219949
- [Background] Morrison CS, Chen PL, Kwok C, Baeten JM, Brown J, Crook AM, Van Damme L, Delany-Moretlwe S, Francis SC, Friedland BA, Hayes RJ, Heffron R, Kapiga S, Karim QA, Karpoff S, Kaul R, McClelland RS, McCormack S, McGrath N, Myer L, Rees H, van der Straten A, Watson-Jones D, van de Wijgert JH, Stalter R, Low N. Hormonal contraception and the risk of HIV acquisition: an individual participant data meta-analysis. PLoS Med. 2015 Jan 22;12(1):e1001778. doi: 10.1371/journal.pmed.1001778. eCollection 2015 Jan. PMID 25612136
- [Background] Govender Y, Avenant C, Verhoog NJ, Ray RM, Grantham NJ, Africander D, Hapgood JP. The injectable-only contraceptive medroxyprogesterone acetate, unlike norethisterone acetate and progesterone, regulates inflammatory genes in endocervical cells via the glucocorticoid receptor. PLoS One. 2014 May 19;9(5):e96497. doi: 10.1371/journal.pone.0096497. eCollection 2014. PMID 24840644
- [Background] Morrison C, Fichorova RN, Mauck C, Chen PL, Kwok C, Chipato T, Salata R, Doncel GF. Cervical inflammation and immunity associated with hormonal contraception, pregnancy, and HIV-1 seroconversion. J Acquir Immune Defic Syndr. 2014 Jun 1;66(2):109-17. doi: 10.1097/QAI.0000000000000103. PMID 24413042
- [Background] Butler AR, Smith JA, Polis CB, Gregson S, Stanton D, Hallett TB. Modelling the global competing risks of a potential interaction between injectable hormonal contraception and HIV risk. AIDS. 2013 Jan 2;27(1):105-113. doi: 10.1097/QAD.0b013e32835a5a52. PMID 23014519
- [Background] Devoize JL, Sztark G, Mehou-Loko A, Foo Cheung L, Joyes B. [Neurological manifestation of multiple cholesterol embolization syndrome: Value of MRI diffusion sequence]. Rev Neurol (Paris). 2013 Nov;169(11):913-6. doi: 10.1016/j.neurol.2012.11.006. Epub 2013 Mar 21. No abstract available. French. PMID 23523018
- [Background] Draper BH, Morroni C, Hoffman M, Smit J, Beksinska M, Hapgood J, Van der Merwe L. Depot medroxyprogesterone versus norethisterone oenanthate for long-acting progestogenic contraception. Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD005214. doi: 10.1002/14651858.CD005214.pub2. PMID 16856087
- [Background] Polis CB, Curtis KM, Hannaford PC, Phillips SJ, Chipato T, Kiarie JN, Westreich DJ, Steyn PS. An updated systematic review of epidemiological evidence on hormonal contraceptive methods and HIV acquisition in women. AIDS. 2016 Nov 13;30(17):2665-2683. doi: 10.1097/QAD.0000000000001228. PMID 27500670